CLINICAL TRIAL: NCT07361250
Title: Evaluation of the Efficacy and Safety of Transcranial Temporal Interference Stimulation (TIS) Targeting the Subthalamic Nucleus (STN) in Parkinson's Disease: A Single-Center, Prospective, Double-Blind, Randomized Controlled Clinical Trial
Brief Title: Subthalamic Nucleus (STN) Targeted Transcranial Temporal Interference Stimulation (TIS) Treats Parkinson's Disease
Acronym: TIS-STN-PD1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tang Zhouping (Other)
Responsible Party: Sponsor-Investigator, Tang Zhouping, Principal Investigator, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202511129
Record Dates: First submitted 2025-12-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Temporal Interference Stimulation; Subthalamic Nucleus (STN)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind trial where participants, investigators administering the intervention, and outcome assessors are blinded. Due to the operation of the Temporal Interference Stimulation device, only the instrument operator administering the experimental stimulation in this experiment is non-blinded. Identical stimulation procedures are used for both groups, with the sham group receiving a non-effective frequency pair.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active TIS stimulation (Experimental): Participants in this group will receive transcranial temporal interference stimulation targeting the subthalamic nucleus using a frequency pair of 2000 Hz and 2130 Hz. Stimulation will be delivered twice daily at the same time for 30 minutes per session over five consecutive days（only once on the 5th day）. Stimulation intensity will be individually titrated starting from a low level and gradually increased to the maximum tolerable level. All treatments will be administered during the participant's medication "on" state.
  Interventions: Device: NervioX-1000
- Sham stimulation (Sham Comparator): Participants in this group will receive sham stimulation using a frequency pair of 2000 Hz and 2000 Hz. Stimulation will be administered twice daily for 30 minutes per session over five consecutive days（only once on the 5th day） during the participant's medication "on" state, with current intensity individually titrated in the same manner as the active group. The sham protocol includes cutaneous sensation simulation during a 30-second ramp-up and ramp-down phase to maintain participant blinding, but does not generate an effective interference field in the deep brain target.
  Interventions: Device: NervioX-1000

INTERVENTIONS:
Device: NervioX-1000 — All participants will receive individualized T1-weighted MRI scans for computational modeling to determine optimized electrode placement and stimulation parameters for transcranial temporal interference stimulation targeting the subthalamic nucleus. The stimulation protocol is designed to generate a focal 130 Hz interference field in the target region while minimizing cortical activation. Parameters including electrode positions and current intensity are customized based on each participant's unique neuroanatomy to ensure precise and tailored neuromodulation.

SUMMARY:
This is a single-center, prospective, double-blind, randomized controlled trial to evaluate the efficacy and safety of transcranial temporal interference stimulation targeting the subthalamic nucleus in patients with Parkinson's disease. It plans to enroll 20 eligible participants who will be randomly assigned in a 1:1 ratio to either the active TIS stimulation group or the sham stimulation group.

DETAILED DESCRIPTION:
Parkinson's disease is a progressive neurodegenerative disorder characterized by motor dysfunction.

Temporal Interference Stimulation (TIS) is a non-invasive deep brain stimulation technique. Its core principle involves placing two pairs of transcranial stimulation electrodes on the scalp surface, each delivering high-frequency currents with slight differences. Since the human cerebral cortex does not respond to high-frequency currents, when these two currents intersect in the deep brain (i.e., the target area), they generate a low-frequency interference wave-similar to tACS-with a frequency equal to the difference between the two currents. This enables selective modulation of deep brain regions while minimizing activation of the superficial cortex. Additionally, a breakthrough aspect of TIS is its ability to flexibly adjust the stimulation target location by modifying electrode positions and current ratios. This makes it highly suitable for future clinical applications in regulating deep brain nuclei and developing personalized diagnosis and treatment plans for Parkinson's disease (PD) patients. The technology offers a non-invasive method to alter neuronal activity in deep brain nuclei and has shown promise in improving PD motor symptoms in prior proof-of-concept studies, thereby providing a potential treatment for PD motor symptoms.

In animal models, TIS has been demonstrated to have the potential to modulate the activity of brain regions closely associated with PD motor symptoms, such as the subthalamic nucleus and globus pallidus. Preliminary clinical studies have shown that TIS stimulation of the unilateral STN in PD patients resulted in alleviation of motor symptoms such as tremor and bradykinesia before and after treatment . A recent exploratory study on TIS stimulation of the right GPi also confirmed that TIS is feasible and safe for alleviating mild PD motor symptoms, particularly bradykinesia and tremor. Compared to the right side, motor symptoms (especially bradykinesia) on the left side showed more significant improvement. PD patients with more severe bradykinesia and tremor before stimulation experienced greater improvement after TIS. Current research findings suggest that TIS has the potential to improve PD motor symptoms. However, in these two studies, some patients did not respond to TIS stimulation. Although preliminary data support the therapeutic potential of TIS for PD motor symptoms, there is still a lack of large-sample, randomized controlled, and systematic studies targeting different brain regions and parameter systems. Therefore, there is an urgent need to conduct standardized clinical trials to evaluate the optimal stimulation parameters, target selection, efficacy persistence, and safety of TIS, providing evidence-based support for its further promotion and application.

This study employs a single-center, prospective, randomized, double-blind, sham-controlled design to evaluate the efficacy and safety of TIS targeting the subthalamic nucleus in Parkinson's disease patients. The study protocol involves structural MRI scanning for all participants to establish individualized computational models, with neuronavigation techniques determining optimal electrode placement. Participants are randomized to either the active stimulation group (using 2000/2130 Hz dual-frequency configuration) or the sham control group (using 2000/2000 Hz configuration). All treatment sessions are conducted during patients' "ON" medication state, administered twice daily for 30 minutes over five consecutive days. Assessment is performed through blinded evaluation by raters unaware of group allocation using standardized scales at predetermined time points. The entire process follows structured data collection and safety monitoring protocols. This study aims to systematically evaluate the therapeutic effects and safety profile of TIS for motor symptoms in Parkinson's disease, providing an evidence base for the clinical application of this novel neuromodulation approach.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older, no gender restriction;
2. Diagnosis of primary Parkinson's disease according to MDS criteria: specifically, the patient must (a) exhibit parkinsonism (bradykinesia + resting tremor/rigidity); (b) not meet any of the MDS absolute exclusion criteria; and (c) meet at least two MDS supportive criteria.
3. Disease duration ≥1 year, stable condition;
4. Hoehn-Yahr stage between 1.5 and 3, with a stable dose of levodopa or other dopaminergic medications for at least 4 weeks, responsive to levodopa-like medications, and no changes to the treatment regimen during the trial;
5. Good compliance, with the patient and family willing to participate in the clinical trial, voluntarily sign the informed consent form, attend regular treatments and follow-ups, and accurately complete evaluation tasks.

Exclusion Criteria:

1. Severe cognitive impairment, resulting in poor compliance due to dementia, and/or inability to sign the informed consent form;
2. History of severe psychiatric disorders, patients with a Hamilton Depression Scale (HAMD) score >24;
3. History of taking antipsychotic drugs, antidepressants, or other medications that may affect dopamine levels;
4. History of seizures within the last year or a family history of epilepsy;
5. Unable to complete MRI scanning (e.g., due to claustrophobia, or having metal implants in the body);
6. Patients with severe heart, liver, or kidney diseases, severe hypertension, and severe orthostatic hypotension that affect their health condition;
7. Patients with severe diabetes or severe cardio-cerebrovascular diseases that affect their health condition;
8. Diagnosed with malignant tumors;
9. Contraindications for non-invasive electrical stimulation, such as intracranial active implants (regardless of whether they are turned on) or passive implants that may affect electrical stimulation treatment, those who have undergone stereotactic deep brain stimulation or neurotomy, or have had any surgical procedures within the last six months that the investigator believes may affect this trial;
10. History of traumatic brain injury;
11. Pregnant women or women planning to become pregnant;
12. Subjects currently participating in other clinical trials or have participated in other clinical research within the last three months without reaching primary endpoints;
13. Patients deemed unsuitable to participate in this clinical study by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Change in Score on Part III (Motor Examination) of the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Baseline (before treatment), immediately after the 1st（day1）, 5th（day3）, and 9th（day5） stimulation sessions (each session lasts for 30 min), and at the two-week and four-week follow-ups after the completion of treatment.
  The motor function of patients was assessed using Part III of the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS-III), which has a total score range of 0 to 132. In this scale, a higher score indicates greater severity of motor symptoms and therefore a worse outcome, with 0 representing no impairment and 132 representing the most severe impairment. Changes in the score reflect the degree of improvement in motor function.

SECONDARY OUTCOMES:
MDS-UPDRS Scale Part I Non-Motor Function Score Changes | Baseline (before treatment), immediately after the 9th（day5） stimulation sessions (each session lasts for 30 min), and at the two-week and four-week follow-ups after the completion of treatment.
  The MDS-UPDRS Scale Part I Non-Motor Function score was used to assess the patient's Cognitive impairment, hallucinations and psychiatric symptoms, depression, apathy, impulse control disorders/dopamine dysregulation syndrome, sleep disorders, pain and other sensory symptoms, and urinary symptoms, with changes in the score reflecting the degree of improvement in those functions. The score for Part I ranges from 0 to 52 points. A higher score indicates greater impairment or more severe non-motor symptoms.
MDS-UPDRS Scale Part II: Activities of Daily Living Score Changes | Baseline (before treatment), immediately after the 9th（day5） stimulation sessions (each session lasts for 30 min), and at the two-week and four-week follow-ups after the completion of treatment.
  The MDS-UPDRS Scale Part II score was used to assess the patient's Activities of Daily Living, with changes in the score reflecting the degree of improvement in daily functions. The score for Part II ranges from 0 to 52 points. A higher score indicates greater impairment in daily activities.
MDS-UPDRS Scale Part IV: Motor Fluctuations, Dyskinesias, and Dystonia Score Changes | Baseline (before treatment), immediately after the 9th（day5） stimulation sessions (each session lasts for 30 min), and at the two-week and four-week follow-ups after the completion of treatment.
  The MDS-UPDRS Scale Part IV score was used to assess the patient's Motor Fluctuations, Dyskinesias, and Dystonia. The score for Part IV ranges from 0 to 24 points. A higher score indicates more severe motor complications caused by long-term levodopa therapy.
Change in Score on the 39-item Parkinson's Disease Questionnaire (PDQ-39) | Baseline (before treatment), immediately after the 9th（day5） stimulation sessions (each session lasts for 30 min), and at the two-week and four-week follow-ups after the completion of treatment.
  The 39-item Parkinson's Disease Questionnaire (PDQ-39) is used to assess the disease-specific health-related quality of life in patients with Parkinson's disease. The summary index score ranges from 0 to 100 points. A higher score indicates a poorer quality of life.
Change in Score on the Hamilton Depression Rating Scale (HAMD) | Baseline (before treatment), immediately after the 9th（day5） stimulation sessions (each session lasts for 30 min), and at the two-week and four-week follow-ups after the completion of treatment.
  Change in Score on the Hamilton Depression Rating Scale (HAMD) is used to evaluate the severity of depressive symptoms. This assessment consists of 17 items with a total score range from 0 to 54 points; a higher score indicates a worse outcome. With common clinical thresholds (e.g., 0-7 = Normal, 8-16 = Mild Depression, 17-23 = Moderate Depression, ≥24 = Severe Depression).
Change in Score on the Hamilton Anxiety Rating Scale (HAMA) | Baseline (before treatment), immediately after the 9th（day5） stimulation sessions (each session lasts for 30 min), and at the two-week and four-week follow-ups after the completion of treatment.
  The Hamilton Anxiety Rating Scale (HAMA) is a 14-item scale to evaluate the severity of anxiety symptoms, where each item is rated on a scale from 0 to 4. The HAMA total score ranges from 0 to 56, with lower scores indicating fewer anxiety symptoms.
Change in Score on the Visual Analog Scale for Fatigue (VAS-Fatigue) | Baseline (before treatment), immediately after the 9th（day5） stimulation sessions (each session lasts for 30 min), and at the two-week and four-week follow-ups after the completion of treatment.
  Visual Analog Scale for Fatigue is used to quantify the subjective intensity of fatigue. The score typically ranges from 0 to 10 cm, where 0 represents "no fatigue" and 10 represents "the worst imaginable fatigue. A higher score indicates greater fatigue severity
Change in Score on the Pittsburgh Sleep Quality Index (PSQI) | Baseline (before treatment), immediately after the 9th（day5） stimulation sessions (each session lasts for 30 min), and at the two-week and four-week follow-ups after the completion of treatment.
  the Pittsburgh Sleep Quality Index (PSQI) is used to assess sleep quality and disturbances over the past month. With changes in the score reflecting the multiple factors of daily function. Each component is scored from 0 to 3. The global PSQI score is the sum of the 7 component scores, ranging from 0 to 21 points. A higher total score indicates poorer sleep quality
Changes in Magnetoencephalography (MEG) | Baseline (before treatment) and immediately after the 9th（day5） stimulation sessions (each session lasts for 30 min).
  Magnetoencephalography (MEG) is a non-invasive, functional neuroimaging technique that measures the magnetic fields generated by the electrical activity of neurons in the brain. It provides direct, real-time (millisecond resolution) information about brain function. With changes in MEG reflecting the brain functional connectivity before and after treatment

OTHER OUTCOMES:
The incidence of SAE | From the first stimulation session until the end of the study follow-up period (each stimulation session lasts for 30 minutes; total study duration including follow-up is 5 weeks). SAEs will be monitored and recorded continuously throughout this period.
  The incidence of SAE
All-cause mortality | 1month after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Zhouping Tang, PhD MD, Principal Investigator — Tongji Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei 450001

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yang C, Xu Y, Du Y, Shen X, Li T, Chen N, Zhu Y, Li L, Huang L, Lu J, Qian Z, Wang Z, Zhou J, Ziemann U, Zhang C, Liu Y. Transcranial temporal interference subthalamic stimulation for treating motor symptoms in Parkinson's disease: A pilot study. Brain Stimul. 2024 Nov-Dec;17(6):1250-1252. doi: 10.1016/j.brs.2024.10.012. Epub 2024 Oct 30. No abstract available. PMID 39486623
- [Result] Violante IR, Alania K, Cassara AM, Neufeld E, Acerbo E, Carron R, Williamson A, Kurtin DL, Rhodes E, Hampshire A, Kuster N, Boyden ES, Pascual-Leone A, Grossman N. Non-invasive temporal interference electrical stimulation of the human hippocampus. Nat Neurosci. 2023 Nov;26(11):1994-2004. doi: 10.1038/s41593-023-01456-8. Epub 2023 Oct 19. Erratum In: Nat Neurosci. 2023 Dec;26(12):2252. doi: 10.1038/s41593-023-01517-y. PMID 37857775
- [Result] Grossman N, Bono D, Dedic N, Kodandaramaiah SB, Rudenko A, Suk HJ, Cassara AM, Neufeld E, Kuster N, Tsai LH, Pascual-Leone A, Boyden ES. Noninvasive Deep Brain Stimulation via Temporally Interfering Electric Fields. Cell. 2017 Jun 1;169(6):1029-1041.e16. doi: 10.1016/j.cell.2017.05.024. PMID 28575667
- See also: Related Info — https://www.nature.com/articles/s41593-023-01456-8